CLINICAL TRIAL: NCT03862833
Title: Phase 1 Dose Escalation of Early Infusion of Zoledronic Acid in Combination With Increasing Low-dose of Interleukin-2 in Order to Expand Vγ9Vδ2 T Cells After T-replete Haplo-identical Allogeneic Stem Cell Transplantation (SCT)
Brief Title: Zoledronic Acid in Combination With Interleukin-2 to Expand Vγ9Vδ2 T Cells After T-replete Haplo-identical Allotransplant
Acronym: HILDEGAZ
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC18_0419
Record Dates: First submitted 2019-02-27; First posted 2019-03-05 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Hematopoietic Stem Cell Transplantation
Keywords: Haplo-SCT; Phase 1; Zoledronic acid; IL-2; g/d T cells
MeSH Terms: interventions — Interleukin-2; Zoledronic Acid

STUDY DESIGN:
Intervention Model Description: a group of patient will received IL2+ zoledronic acid a group of patient will not received IL2+ zoledronic acid
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): Zoledronic acid and IL-2 Zoledronic acid: 4 mg
  Three IL2 levels will be tested:
  Level 1: 2 millions UI/Infusion Level 2: 4 millions UI/Infusion Level 3: 6 millions UI/Infusion
  Interventions: Drug: IL2; Drug: Zoledronic Acid
- control group (No Intervention): no experimental treatment

INTERVENTIONS:
Drug: IL2 — Three IL2 levels will be tested:
  Level 1: 2 millions UI/Infusion Level 2: 4 millions UI/Infusion Level 3: 6 millions UI/Infusion 4 weeks, 5 days per week from day + 15 post graft to day + 40
  Arms: experimental group
Drug: Zoledronic Acid — 4 mg at day +15 post graft
  Arms: experimental group

SUMMARY:
Patients receiving haplo-SCT are at high-risk of relapse. Vγ9Vδ2 T cells exhibit is a well-known population able to exert cytotoxicity toward a large range of tumor in vitro or in vivo. Activating and expanding Vγ9Vδ2 T cells early after haplo-SCT by using a combination of Zoledronic acid and low-dose interleukine (IL) -2 may be of benefit for patients by reducing incidence of relapse. The optimal dose of IL-2 to use remains to be determined.

This will be a Phase 1 3+3 escalation study. Three to 15 patients are planned. It will be proposed to Patients who refuse to participate to have samples collected until day +70 to study immune and gamma/delta T cells reconstitutions after haplo-transplant.

DETAILED DESCRIPTION:
Zoledronic acid will be administered as a single dose according to marketing and regulatory authorization at the dose of 4 mg over 15 min intravenously at day+15 post-transplant. Zoledronic acid infusion must be stopped in case of grade 3/4 adverse events during infusion.

IL-2 will be administered at a unique low-dose level 5 days per week for 4 consecutive weeks from Monday to Friday subcutaneously . IL-2 has already marketing authorization for various indications.

Three IL2 levels will be tested:

Level 1: 2 millions UI/Infusion Level 2: 4 millions UI/Infusion Level 3: 6 millions UI/Infusion Zoledronic acid and IL2 have to start at day+15 if it is a Monday or the first Monday following day+15 in order to avoid administration on week-end.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-70 years old
* Patients with a hematological disease eligible for a haplo-SCT using the Baltimore regimen as conditioning regimen (Luznik, BBMT, 2008) (See 5.1.2)
* Patients with no HLA matched sibling or unrelated donors
* ECOG <=2
* Signed informed consent
* Patient affiliated to or beneficiary of the National Health Service
* Patients previously transplanted are eligible to the study

Exclusion Criteria:

* Patients with a HLA matched sibling or unrelated donor
* Active uncontrolled infections
* HIV positive, active Hepatitis B or C
* Childbearing or child-breastfeading women
* Women or men without effective contraceptive barrier if needed
* Left ventricular ejection fraction < 50% with no previous severe cardiopathy
* Respiratory insufficiency defined as DLCO <40% of the corrected value
* Creatinine clearance <50 ml/min
* Serum bilirubin >2.5 or transaminases >5 fold of normal value except if due to the hematological disease
* Previous or concurrent second malignancy except for adequately treated basal cell carcinoma of the skin, curatively treated in situ carcinoma of the cervix, curatively treated solid cancer, with no evidence of disease for at least 2 years
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule
* Participation at the same time in another study in which investigational drugs are used
* Absence of written informed consent
* Contra-indication to Zoledronic acid: known hypersensitivity to Zoledronic acid or other bisphosphonate or Zoledronic acid formulation (excipients)
* Recent or programmed dental care
* Contra-indication to IL-2: known hypersensitivity to IL-2 or IL-2 formulation (excipients)
* No previous ou current use of zoledronic acid

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-05-07 (Actual); Primary Completion 2023-08-29 (Actual); Study Completion 2023-08-29 (Actual)

PRIMARY OUTCOMES:
determine the maximum tolerated dose (MTD) of early administration of increasing doses of low-dose IL-2 in combination with a fixed dose of Zoledronic acid after haplo-SCT | 28 days after the last injection of IL2
  A dose-limiting toxicity (DLT) will be defined as:
  * non-hematological toxicity of grade 4, including grade 4 acute GVHD 4.
  * non-hematological toxicity of grade 3 non-reversible for > 7 days or reappearance of the same grade 3 after reintroduction of IL2 in case of return to at least one grade 1.
  * an acute GVHD grade 2-3 for > 7 days or reappearance of GVHD grade 2-3 acute GVHD after reintroduction of IL2 if at least grade 1 acute GVHD is restored.
  * a reappearance of a grade 3/4 IL2 allergic reaction after reintroduction of IL2 in the event of a return to at least grade 1 after the occurrence of an allergic reaction of grade 3/4 IL2 when of the administration.
  * grade 4 pancytopenia with hypocellular bone marrow (no disease detection) for > 4 weeks after the last administration of IL2.

SECONDARY OUTCOMES:
Engraftment | day 30, 60,90/100, 6 months and 1 year post-transplant
  Concentration of sustained neutrophil recovery (>500 Giga/L) with full or mixed donor chimerism documentation
Chimerism (mixed, full or uncompleted) | day 30, 60,90/100, 6 months and 1 year post-transplant
  Evaluation of CD3+ T-cell chimerism
overall survival | last patient follow up : 36 months
  the time from day 0 of allo-SCT to death or last follow-up for surviving patients
disease-free survival | last patient follow up : 36 months
  time from day 0 of allo-SCT to time without evidence of relapse or disease progression censored at the date of death or last follow-up.
relapse rate | last patient follow up : 36 months
  any event related to re-occurrence of the disease.
Non relapse mortality | day 100 post transplant and one year post-transplant
  death from any cause without previous relapse or progression
Incidence of acute GVHD | day 100 post transplant one year post-transplant
  Acute GVHD: Harris AC, Young R, Devine S, Hogan WJ, Ayuk F, Bunworasate U, et al. International, Multicenter Standardization of Acute Graft-versus-Host Disease Clinical Data Collection: A Report from the Mount Sinai Acute GVHD International Consortium. Biol Blood Marrow Transplant. 2016 Jan;22(1):4-10.
Hematologic and immune reconstitutions post-transplant | before the graft and at days 15, 22, 29, 36, 45, 70
  median time for neutrophils recovery (first day with >0.5 Giga/L for three consecutive days) and platelets recovery >20, 50 and 100 Giga/L; T CD3, CD4, CD8, NK, B, Tregs, g/d T cells
Complete remission (CR) rate for lymphoma patients | day 100 post transplant
  Cheson criteria
g/d T cells detection after haplo-SCT | before the graft and at days 15, 22, 29, 36, 45, 70
  Evaluation of T CD3, CD4, CD8, NK, B, Tregs, g/d T cells
Perturbation of ionic metabolism | before the graft and at days 15, 22, 29, 36, 45, 70
  Evaluation of Vitamin D, Ca, Ph, Na, K, serum creatinine, bilirubin (direct and total), alkaline phosphatase, gammaGT, ALAT, ASAT
Detection of dysthyroid disease | before the graft and at day 70
  Dosage of T3 T4 TSH
Incidence of acute and chronic GVHD | one year post-transplant
  Chronic GVHD: Filipovich AH, Weisdorf D, Pavletic S, Socie G, Wingard JR, Lee SJ, et al. National Institutes of Health consensus development project on criteria for clinical trials in chronic graft-versus-host disease: I. Diagnosis and staging working group report. Biol Blood Marrow Transplant. 2005 Dec;11(12):945-56.

CONTACTS AND LOCATIONS:
Locations (1):
- Nantes Uh, Nantes, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jullien M, Guillaume T, Le Bourgeois A, Peterlin P, Garnier A, Eveillard M, Le Bris Y, Bouzy S, Tessoulin B, Gastinne T, Dubruille V, Touzeau C, Mahe B, Blin N, Lok A, Vantyghem S, Sortais C, Antier C, Moreau P, Scotet E, Bene MC, Chevallier P. Phase I study of zoledronic acid combined with escalated doses of interleukine-2 for early in vivo generation of Vgamma9Vdelta2 T-cells after haploidentical stem cell transplant with posttransplant cyclophosphamide. Am J Hematol. 2024 Mar;99(3):350-359. doi: 10.1002/ajh.27191. Epub 2024 Jan 2. PMID 38165016